CLINICAL TRIAL: NCT00127634
Title: A Pivotal Long-Term, Open-Label, Parallel Study of the Efficacy and Safety of Human Insulin Inhalation Powder in Patients With Type 1 Diabetes Mellitus
Brief Title: Study of Human Insulin Inhalation Powder in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6120; H7U-MC-IDAH
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Human Insulin Inhalation Powder; Drug: Insulin Glargine
- 2 (Active Comparator)
  Interventions: Drug: Injectable Insulin; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Human Insulin Inhalation Powder — patient specific dose, inhaled, before meals, 24 months, up to 36 months
  Other Names: LY041001
  Arms: 1
Drug: Injectable Insulin — patient specific dose, injectable, before meals, 24 months, up to 36 months.
  Arms: 2
Drug: Insulin Glargine — patient specific dose, injectable, as needed, 24 months up to 36 months

SUMMARY:
This is a phase 3, open-label, randomized study to evaluate the safety and efficacy of the Lilly/Alkermes inhaled insulin system compared to injected pre-meal insulin in non-smoking patients with type 1 diabetes. Patients will be treated for 24 months with a 2-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Non smoker
* Normal lung function

Exclusion Criteria:

* Significant pulmonary, hepatic, or renal disease
* Severe congestive heart failure
* Active malignancy
* Systemic glucocorticoid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2005-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To assess change in baseline to endpoint in HbA1c in type 1 diabetic patients. | 24 months

SECONDARY OUTCOMES:
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to FEV1, FVC, and total lung capacity (TLC), and diffusing capacity of the lung for carbon monoxide (DLCO). | 24 months
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to safety as assessed by insulin antibody binding levels, adverse events, and episodes of hypoglycemia | 24 months
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to safety using serial HRCT scans of the chest | 24 months
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to safety as assessed by Six-Minute Walk Test with the Borg CR10 scale to access perceived exertion. | 24 months
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to proportion of patients who achieve or maintain an HbA1c < 7.0 %. | 24 months
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to insulin dose requirements ( total, preprandial, and basal insulin) | 24 months
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to Patient reported questionnaires. | 24 months
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to resource utilization | 24 months
To assess inhaler reliability in patients randomized to treatment with Human Insulin Inhalation Powder. | throughout the study
To explore differences in cough and other pulmonary symptoms in patients treated with Human Insulin Inhalation Powder or preprandial injectable insulin using the Pulmonary Symptom Questionnaire. | months 32, 38, 40 and ED visits
To compare preprandial Human Insulin Inhalation Powder with preprandial injectable insulin in patients with type 1 diabetes with respect to glycemic control as assessed by the 8-point self-monitored blood glucose profiles | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (61):
- United States (35):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Walnut Creek, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Largo, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Plainfield, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flushing, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Success, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Hyde Park, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medford, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Downingtown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sellersville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Belgium (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corunna, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niagara Falls, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peterborough, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarnia, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb, Croatia
- Hungary (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eger
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyula
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kecskemét
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Szeged
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Dehli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Noida

REFERENCES:
- [Derived] Garg SK, Mathieu C, Rais N, Gao H, Tobian JA, Gates JR, Ferguson JA, Webb DM, Berclaz PY. Two-year efficacy and safety of AIR inhaled insulin in patients with type 1 diabetes: An open-label randomized controlled trial. Diabetes Technol Ther. 2009 Sep;11 Suppl 2:S5-S16. doi: 10.1089/dia.2009.0040. PMID 19772449
- See also: Lilly CSR synopsis — https://www.lilly.com/clinical-study-report-csr-synopses